CLINICAL TRIAL: NCT02319382
Title: High Resolution PET Imaging of Microglial Activation in Parkinson's Disease (PD) With a New Tracer [18F]DPA-714
Brief Title: Measure of Microglial Activation in the Brain of Parkinson Disease Patients With PET
Acronym: INFLAPARK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: France Parkinson Association (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: P091202
Record Dates: First submitted 2014-11-18; First posted 2014-12-18 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-07

CONDITIONS: Parkinson's Disease With LRRK2 Mutation; Healthy Controls; Parkinson's Disease Without LRRK2 Mutation
Keywords: Parkinson Disease; [18F]DPA-714; Positron emission tomography (PET); Neuroinflammation
MeSH Terms: conditions — Parkinson Disease; Neuroinflammatory Diseases | interventions — 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 2 markers: 18F-DPA-714 and 11C-PE2I (Experimental): PET with the tracer [18F]DPA-714 and second PET with the tracer [11C]-PE2I. [18F]DPA-714 is a new marker. It allows the macroscopic visualization of active microglia in the brain. [11C]-PE2I allow measures dopaminergic neuronal loss.
  Interventions: Radiation: PET with the tracer 18F-DPA-714; Radiation: PET with the tracer 11C-PE2I; Other: MRI

INTERVENTIONS:
Radiation: PET with the tracer 18F-DPA-714
Radiation: PET with the tracer 11C-PE2I
Other: MRI — Magnetic field

SUMMARY:
There is accumulating evidence suggesting that inflammatory processes, through microglial activation, would play a key role in the neurodegenerative process of Parkinson's disease (PD). It is considered that microglial activation would be part of self-propelling cycle of neuroinflammation that fuels the progressive dopaminergic neurodegeneration. It is however hard to evidence microglial activation in vivo, especially in the substantia nigra: first, the investigators need very high resolution imaging tools and then, the only ligand available to date, 11C-PK11195, has a low sensitivity and specificity and provided heterogeneous results.

18F-DPA-714 is a new PET ligand which labels microglial cells. The investigators aim to explore the topography and intensity of microglial activation in several different groups of PD patients: 1) de novo, drug-naïve subjects (n = 6); 2) non-fluctuating treated patients ("honeymoon") (n = 10); 3) advanced drug-responsive patients motor fluctuations (wearing-off or dyskinesia) (n = 6); 4) patients with LRRK2 gene mutation (n = 6); and 5) related to healthy patients carriers of the mutation LRRK2(n = 6). PET imaging will be performed with a new generation tomography having a very high resolution.

This study might reveal significant neuroinflammatory process in the midbrain of PD patients and will determine if such process is present in both sporadic and genetic forms of PD. The results of this study might provide a new biomarker of disease pathological progression and help as identifying subjects who might most benefit from a specific anti-inflammatory drug.

ELIGIBILITY:
Inclusion Criteria:

For all subjects:

The subject is an out-patient aged 18 years or above Active affiliation to national health insurance system Signed informed consent to participate in the study

Additional criteria depending on the group under study:

Group 1:

Parkinson disease diagnosed for less than 18 months and no treatment Age at disease over 40 years

Group 2:

Disease Parkinson diagnosed for less than 36 months and treated by L-Dopa or /and dopaminergic agonist No motor fluctuation Age at disease over 40 years

Group 3:

Parkinson disease diagnosed for more than 3 years Age at disease over 40 years Motor fluctuations for more than 6 months (dyskinesia or wearing off )

Group 4:

Parkinson disease LRRK2 mutation proved by genetic analysis

Group 5:

LRRK2 mutation proved by genetic analysis No evidence of Parkinson disease attested by a Unified Parkinson's Disease Rating Scale (UPDRS) score of 0 or1

Group 6:

No evidence of Parkinson disease attested by a UPDRS score of 0 or1

Exclusion Criteria:

For all subjects:

Contraindication for MRI Anti-inflammation treatment for more 50 days during previous year or for more 7 days during previous month Pregnancy or lactating Legal incapacity or limited legal capacity Beneficiary of AME

Additional criteria depending on the group under study:

Group 1:

Atypical parkinsonism Other neurological diseases or known brain lesion

Group 2:

Atypical parkinsonian syndrome

Group 3:

Atypical parkinsonian syndrome Resistance to treatment (benefit of treatment estimated to less than 30%) Other neurological diseases or known brain lesion

Groups 4 and 5:

Other neurological diseases or known brain lesion

Group 6:

Previous neurological or psychiatry diseases or known brain lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2012-06; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Accumulation of [18F]DPA-714 in the midbrain assessed through PET | Inclusion visit

CONTACTS AND LOCATIONS:
Overall Officials: Philippe REMY, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Orsay Hospital, Orsay, France

REFERENCES:
- [Derived] Peyronneau MA, Kuhnast B, Nguyen DL, Jego B, Sayet G, Caille F, Lavisse S, Gervais P, Stankoff B, Sarazin M, Remy P, Bouilleret V, Leroy C, Bottlaender M. [18F]DPA-714: Effect of co-medications, age, sex, BMI and TSPO polymorphism on the human plasma input function. Eur J Nucl Med Mol Imaging. 2023 Sep;50(11):3251-3264. doi: 10.1007/s00259-023-06286-1. Epub 2023 Jun 9. PMID 37291448
- [Derived] Ricigliano VAG, Louapre C, Poirion E, Colombi A, Yazdan Panah A, Lazzarotto A, Morena E, Martin E, Bottlaender M, Bodini B, Seilhean D, Stankoff B. Imaging Characteristics of Choroid Plexuses in Presymptomatic Multiple Sclerosis: A Retrospective Study. Neurol Neuroimmunol Neuroinflamm. 2022 Oct 13;9(6):e200026. doi: 10.1212/NXI.0000000000200026. Print 2022 Nov. PMID 36229188
- [Derived] Lavisse S, Goutal S, Wimberley C, Tonietto M, Bottlaender M, Gervais P, Kuhnast B, Peyronneau MA, Barret O, Lagarde J, Sarazin M, Hantraye P, Thiriez C, Remy P. Increased microglial activation in patients with Parkinson disease using [18F]-DPA714 TSPO PET imaging. Parkinsonism Relat Disord. 2021 Jan;82:29-36. doi: 10.1016/j.parkreldis.2020.11.011. Epub 2020 Nov 17. PMID 33242662